CLINICAL TRIAL: NCT06133725
Title: Transversus Abdominis Plane Block Combined With Rectus Sheath Block Versus Erector Spinae Plane Block for Postoperative Analgesia After Laparoscopic Liver Resection
Brief Title: TAPB Combined With RSB Versus ESPB for Postoperative Analgesia After Laparoscopic Liver Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhangyi (Other)
Responsible Party: Sponsor-Investigator, Zhangyi, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: TJ-IRB20230951
Record Dates: First submitted 2023-10-23; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Laparoscopic Hepatectomy; Nerve Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB (Experimental): erector spinae plane block
  Interventions: Procedure: erector spinae plane block
- TAPB&RSB (Active Comparator): transversus abdominis plane block combined with rectus sheath block
  Interventions: Procedure: erector spinae plane block

INTERVENTIONS:
Procedure: erector spinae plane block — The experimental group received ultrasound-guided erector spinae plane block, and bilateral erector spinae plane block was performed at T7 segment with 20ml 0.375% ropivacaine on each side.While the control group received ultrasound-guided transversus abdominis plane block combined with rectus sheath block, which will be performed under the costal margin with 10ml 0.375% ropivacaine for bilateral transversus abdominis plane block and 10ml 0.375% ropivacaine for bilateral rectus sheath block.
  Other Names: transversus abdominis plane block combined with rectus sheath block

SUMMARY:
Postoperative pain after laparoscopic hepatectomy is composed of multiple factors, and the peak pain of postoperative pain mainly occurs within the first 24 hours, so it is particularly important to find an appropriate analgesic method. Transversus abdominis plane block (TAPB) and Rectus sheath blocks (RSB) are widely used in abdominal surgery, but too deep a needle tip during RSB may puncture abdominal organs. TAPB and RSB can only provide somatic analgesia, but lack visceral analgesia. Recently, Erector spinae plane block (ESPB) has been used in some studies for analgesia after abdominal surgery. The purpose of this study is to compare the analgesic effect and postoperative recovery effect of erector spinae plane block and transverse abdominis plane block combined with rectus sheath block in patients undergoing laparoscopic hepatectomy. Therefore, this study has important clinical implications.

DETAILED DESCRIPTION:
In a double-blind randomized controlled study, researchers randomized 60 patients undergoing laparoscopic hepatectomy to TAPB combined with RSB or ESPB, with both groups receiving additional standardized treatment, including multimodal analgesia. The main outcome was the consumption of morphine within 24 hours after surgery. Secondary outcomes included the number of rescue analgesia at 1h, 2h, 4h, 8h and 24 hours after surgery, VAS scores in resting and coughing at 1h, 2h, 4h, 8h and 24h after surgery, CVP values at 5, 10, 15 and 30min after nerve block, QoR-15 patient questionnaire scores before and 24h after surgery, and postoperative liver function (the percentage increase of AST and ALT compare with preoperative), postoperative complications and discharge time.

ELIGIBILITY:
Inclusion Criteria:

1. ASA grades I-II;
2. Age 18~70 years old;
3. BMI 19～28kg/m2;
4. Patients undergoing elective laparoscopic partial liver resection;

Exclusion Criteria:

1. The nerve block cannot be performed, such as skin infection at the puncture site;
2. Daily using the opioid analgesics or have a history of opioid abuse;
3. Allergy or a history of drug allergy to any of the drugs used in the study;
4. Patients have cognitive impairment, mental or neurological diseases, motor or sensory deficits;
5. Coagulation disorders;
6. Severe lung, heart, liver, or kidney dysfunction;
7. Participating in other clinical trials within 3 months before being included in this study;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
The dose of morphine used | 24 hours after surgery
  dosage of analgesic pump

SECONDARY OUTCOMES:
The dose of morphine used | 1hour, 2hours, 4hours and 8hours after surgery
  dosage of analgesic pump
The number of rescue analgesia | 1hour, 2hours, 4hours, 8hours and 24hours after surgery
  times of rescue analgesia
Visual analogue scale scores in resting and coughing state | 1hour, 2hours, 4hours, 8hours and 24hours after surgery
  Visual analogue scale (VAS): a 100 mm transverse line with 0mm at one end of the line indicates no pain, 100mm at the other end indicates severe pain and the middle part shows different levels of pain.
The value of central venous pressure | 5min, 10min, 15min and 30min after nerve block
  ultrasound-guided internal jugular vein catheterization connected with transducer
QoR-15 scores | before and 24h after surgery
  The QOR-15 scale was scored from 0 (very poor QoR) to 150 (excellent QoR). A higher score indicates a better patient status.
Quantitative assessment of liver function | before and 1days, 3days after surgery
  The levels of plasma liver function markers AST and ALT before and after liver resection.
Postoperative Complications | 2hours, 4hours, 8hours and 24hours after surgery
  Including nausea, vomiting, pruritus, dizziness, headache, constipation, urinary retention, respiratory depression and so on.
Recovery time nodes | follow up patients for an average of half a month
  drainage tube removal time, offbed activity, or postoperative hospital stay, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu M, Mo X, Zhan R, Wang H, Zhao Y, Zhang Y. Erector spinae plane block versus transversus abdominis plane block with rectus sheath block for postoperative analgesia in laparoscopic hepatectomy: a randomized clinical trial. BMC Anesthesiol. 2025 Apr 9;25(1):162. doi: 10.1186/s12871-025-03031-z. PMID 40205560

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT06133725/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT06133725/ICF_001.pdf